CLINICAL TRIAL: NCT03585959
Title: A Post-market Feasibility Study Evaluating Location Accuracy Using the superDimension™ Navigation System Version 7.2 With Fluoroscopic Navigation Technology in Subjects Undergoing Lung Lesion Biopsy
Brief Title: superDimension™ Navigation System Version 7.2 With Fluoroscopic Navigation Technology
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic - MITG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: MDT18004ILSFNV
Record Dates: First submitted 2018-06-21; First posted 2018-07-13 (Actual); Results first posted 2020-04-07 (Actual); Last update posted 2020-04-29 (Actual); Status verified 2020-04

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Fluoroscopic Navigation Arm (Experimental): An Electromagnetic navigation bronchoscopy (ENB) system which provides enhanced three-dimensional fluoroscopy to improve lesion visibility and to compensate for CT-to-body divergence, with an integrated real-time local registration feature allowing the operator to update the catheter position relative to the target during the procedure.
  Interventions: Device: superDimension™ Navigation System Version 7.2

INTERVENTIONS:
Device: superDimension™ Navigation System Version 7.2 — superDimension™ Navigation System Version 7.2 with Fluoroscopic Navigation Technology in subjects undergoing lung lesion biopsy

SUMMARY:
The purpose of this investigation is to confirm the clinical accuracy of the superDimension™ Navigation System Version 7.2 with Fluoroscopic Navigation Technology.

DETAILED DESCRIPTION:
The primary objective of this post-market feasibility study is to confirm the location accuracy of the local registration feature of the superDimension™ Navigation System Version 7.2 in subjects undergoing lung lesion biopsy.

ELIGIBILITY:
Inclusion Criteria:

1. Subject presents with lung lesion(s) 10 mm or greater in diameter amenable to evaluation by ENB at the time of evaluation
2. Lesion is intended to be biopsied by the participating investigator
3. Subject is willing and able to provide informed consent to participate in the study
4. Subject is a candidate for an elective ENB procedure
5. Subject is over the age of 18

Exclusion Criteria:

1. Central lesions that are visible endobronchially or could be reached by a flexible bronchoscope or endobronchial ultrasound (EBUS) without the utilization of ENB
2. Lesions within 10 mm of the diaphragm
3. The subject is unable or unwilling to comply with study follow-up schedule
4. The subject has participated in an investigational drug or device research study within 30 days of enrollment that would interfere with this study
5. Female subjects who are pregnant or nursing as determined by standard site practices

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2018-08-03 (Actual); Primary Completion 2019-02-13 (Actual); Study Completion 2019-02-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael A. Pritchett, DO MPH, Principal Investigator — FirstHealth Moore Regional Hospital; Krishnendu Bhadra, MD, Principal Investigator — CHI Memorial Medical Group
Locations (2):
- United States (2):
  - FirstHealth Moore Regional Hospital, Pinehurst, North Carolina
  - CHI Memorial Medical Group, Chattanooga, Tennessee

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Fluoroscopic Navigation Arm
Started | 50
Completed | 47
Not Completed | 3
Not completed — Physician Decision | 1
Not completed — Unsuccessful Procedure | 2

BASELINE CHARACTERISTICS:
Population: All enrolled subjects were underwent baseline analysis.
Arm/Group | Fluoroscopic Navigation Arm
Number analyzed (Participants) | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 38
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.8 (7.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35
  Male | 15
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 43
  Black of African American | 5
  American Indian or Alaska Native | 2
Region of Enrollment [Number; unit: participants]
  United States | 50
Medical History [Number; unit: participants]
  Chronic Obstructive Pulmonary Disease (COPD) | 31
  Tobacco Use | 44
Lesion Characteristics [Number; unit: lesion] — Population: Lesion data is only available in subjects with local registration attempted.
  lesion
    Lesion < 20 mm: number analyzed (Participants) | 49
    Lesion < 20 mm | 30
    Upper Lobe Location: number analyzed (Participants) | 49
    Upper Lobe Location | 32
    Pure to mostly solid (Suzuki Class 5 or 6): number analyzed (Participants) | 49
    Pure to mostly solid (Suzuki Class 5 or 6) | 49
    Bronchus Sign Present on CT: number analyzed (Participants) | 49
    Bronchus Sign Present on CT | 26

OUTCOME MEASURES:

1. Primary Outcome: Confirm the Location Accuracy of the Local Registration Feature
Description: The Primary Endpoint is the measured ability of the superDimension™ Navigation System v7.2 with Fluoroscopic Navigation Technology to place the center of the virtual navigation target (green ball) on the intended target lesion as confirmed by cone-beam computed tomography (CBCT).
  The primary endpoint was evaluated in technically successful cases (those with local registration complete) and calculated as the percentage of cases in which the virtual target was correctly placed to overlap the target lesion, as confirmed by CBCT. The percent overlap was calculated in three dimensions (X, Y, and Z coordinates). Any case with more than 0% overlap was considered a primary endpoint success.
Time Frame: day of procedure
Population: 47 cases were technically successful. From 47 cases, 4 couldn't be analyzed due to inadequate video recording. From 43 cases, 2 cases only had data from FNAV/CBCT 1 (Before Correction of Catheter Location) and 2 cases only had data from FNAV/CBCT 2 (After Correction of Catheter Location) resulting in 41 evaluable subjects per FNAV/CBCT group.
Measure: Count of Participants; unit: Participants
Arm/Group | Fluoroscopic Navigation Arm
Number analyzed (Participants) | 47
Participants
  All Technically Successful Cases, FNAV/CBCT 1: Target overlap achieved | 28
  All Technically Successful Cases, FNAV/CBCT 1: Target overlap not achieved | 19
  All Technically Successful Cases, FNAV/CBCT 2: Target overlap achieved | 39
  All Technically Successful Cases, FNAV/CBCT 2: Target overlap not achieved | 8
  All Evaluable Cases, FNAV/CBCT 1: number analyzed (Participants) | 41
  All Evaluable Cases, FNAV/CBCT 1: Target overlap achieved | 28
  All Evaluable Cases, FNAV/CBCT 1: Target overlap not achieved | 13
  All Evaluable Cases, FNAV/CBCT 2: number analyzed (Participants) | 41
  All Evaluable Cases, FNAV/CBCT 2: Target overlap achieved | 39
  All Evaluable Cases, FNAV/CBCT 2: Target overlap not achieved | 2

2. Secondary Outcome: Number of Cases That Are Technically Successful (Successful Completion of Local Registration)
Description: Technical success was defined as successful completion of local registration utilizing fluoroscopic navigation technology.
Time Frame: day of procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Fluoroscopic Navigation Arm
Number analyzed (Participants) | 49
Participants | 47

3. Secondary Outcome: Number of Cases That Are Not Technically Successful (Local Registration Not Complete)
Description: By device design, if the local registration algorithm determines that the correction distance is greater than 3.0 cm the location of the virtual target will not be updated. These cases are not considered technically successful according to the clinical study definitions, even though the device performed as designed.
Time Frame: day of procedure
Population: 2 of 49 cases did not complete local registration
Measure: Count of Participants; unit: Participants
Arm/Group | Fluoroscopic Navigation Arm
Number analyzed (Participants) | 2
Participants | 2

4. Secondary Outcome: Investigator Confirmation That the Catheter is in an "Adequate Periprocedural Location" Using the Electromagnetic Navigation Bronchoscopy (ENB) Technology.
Description: Investigator confirmation that the catheter was in an "adequate periprocedural location" (the location of the extended working channel when the proceduralist made the decision that placement was adequate and clinically acceptable to proceed with tissue sampling). Adequate periprocedural location is reported with use of local registration.
Time Frame: day of procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Fluoroscopic Navigation Arm
Number analyzed (Participants) | 49
Participants | 47

5. Secondary Outcome: Total Procedure Time
Description: Total time from the first entry of the bronchoscope to the final removal of the bronchoscope. This includes all study-specific fluoroscopy and CBCT steps which would not normally occur in standard practice
Time Frame: day of procedure
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Fluoroscopic Navigation Arm
Number analyzed (Participants) | 49
minutes | 65.3 (22.4)

6. Secondary Outcome: ENB Procedure Time
Description: ENB procedure time captured in the electronic data capture database being utilized for the study defined as the total time from the first entry of the extended working channel or locatable guide until the last exit of the extended working channel. This includes all study-specific fluoroscopy and CBCT steps which would not normally occur in standard practice
Time Frame: day of procedure
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Fluoroscopic Navigation Arm
Number analyzed (Participants) | 49
Minutes | 54.3 (20.5)

7. Secondary Outcome: Total Fluoroscopy Time
Description: Total fluoroscopy time captured in the electronic data capture database being utilized for the study was determined to not be clinically relevant. Instead, the fluoroscopic navigation time is presented. Fluoroscopic Navigation Time: Two sweeps pooled. Encompasses c-arm sweep, target marking, and algorithm computational time, inclusive of the initiation of the local registration applet to the time the updated catheter location was ready and on screen (not including CBCT), as measured by the system software
Time Frame: day of procedure
Population: Four cases were considered technically successful but could not be analyzed due to inadequate video recording and an additional four technically successful cases had data from only FNAV/CBCT 1 (n=2) or only FNAV/CBCT 2 (n=2), resulting in evaluable datasets of 41 subjects per FNAV/CBCT group.
Measure: Median (Full Range); unit: Minutes
Units Other Than Participants: Local Registrations
Arm/Group | Fluoroscopic Navigation Arm
Number analyzed (Participants) | 41
Number analyzed (Local Registrations) | 81
Minutes | 3.8 [0.2 to 7.9]

8. Secondary Outcome: Adequacy of the ENB-aided Tissue Sample
Description: Adequacy of the ENB-aided tissue sample for rapid on-site evaluation (ROSE) of cytologic samples by pathology (when applicable). This will be captured in the electronic data capture database.ROSE results could be reported as "Benign", "Inconclusive", "Malignant", "Inadequate Tissue for ROSE", or "N/A". If all ROSE diagnoses were report as "Inadequate Tissue for ROSE", for a participant, then the case was considered as "Inadequate Tissue".
Time Frame: Based on final pathology results of the ENB-aided biopsy sample collected day of procedure
Population: ROSE was attempted in 49/49 cases.
Measure: Count of Participants; unit: Participants
Arm/Group | Fluoroscopic Navigation Arm
Number analyzed (Participants) | 49
Participants | 49

9. Secondary Outcome: Histopathological Call Based on ROSE of the ENB-aided Tissue Sample (When Applicable)
Description: Histopathological call based on ROSE of the ENB-aided tissue sample (when applicable) captured in the electronic data capture database being utilized for the study. Only malignant results are presented, as adequate follow-up to confirm the benign/inconclusive results was not part of the study design.
Time Frame: day of procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Fluoroscopic Navigation Arm
Number analyzed (Participants) | 49
Participants
  Malignant | 26
  Other | 23

10. Secondary Outcome: Final Pathology Results of the ENB-aided Tissue Sample
Description: Final pathology results of the ENB-aided tissue sample captured in the electronic data capture database being utilized for the study. Only malignant results are presented, as adequate follow-up to confirm the benign/inconclusive results was not part of the study design.
Time Frame: Based on final pathology results of the ENB-aided biopsy sample collected day of procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Fluoroscopic Navigation Arm
Number analyzed (Participants) | 49
Participants
  Malignant | 30
  Other | 19

11. Secondary Outcome: Biopsy Tools Used
Description: Biopsy tools used was captured in the electronic data capture database being utilized for the study on all subjects with local registration attempted. If subject use same tool more than once, only counts once.
Time Frame: day of procedure
Measure: Number; unit: tool use
Arm/Group | Fluoroscopic Navigation Arm
Number analyzed (Participants) | 49
tool use
  Aspiration Needle | 42
  Biopsy Forceps | 33
  GenCut Core Biopsy Tool | 10
  Cytology Brush | 49
  superDimension triple needle cytology brush | 2
  superDimension needle-tipped cytology brush | 2
  Bronchoalveolar lavage/washing | 30

12. Secondary Outcome: Tool Order
Description: Tool order analysis reports the number of times that a tool was used first in a patient.
Time Frame: day of procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Fluoroscopic Navigation Arm
Number analyzed (Participants) | 49
Participants
  Aspirating needle | 26
  Cytology brush | 23

13. Secondary Outcome: Number of Tool Pases
Description: An analysis of the number of passes for each tool was planned, but it was determined that it wouldn't be clinically meaningful to go into that level of detail for the analysis and instead focused on the number of passes for only the first tool used.
Time Frame: day of procedure
Measure: Mean (Standard Deviation); unit: passes
Arm/Group | Fluoroscopic Navigation Arm
Number analyzed (Participants) | 49
passes
  Arcpoint pulmonary needle | 6 (4.2)
  Aspirating needle, superDimension | 9 (2.8)
  Cytology brush, non-superDimension | 2 (0)
  Cytology brush, superDimension | 4 (1.8)

14. Secondary Outcome: Diagnoses for Each Tool Based on ROSE of the ENB-aided Sample
Description: The "tool-specific accuracy for malignancy" is calculated out of only the malignant cases using that tool. Only malignant results are presented, as adequate follow-up to confirm the benign/inconclusive results was not a part of the study design.
Time Frame: Based on ROSE results of the ENB-aided biopsy sample collected day of procedure
Population: Patients with overall malignant results by ROSE (26/49 cases). The number analyzed varies by tool based on the number of cases which used each tool. More than one tool could be used per case. Bronchoalveolar Lavage is not applicable for ROSE.
Measure: Number; unit: participants
Arm/Group | Fluoroscopic Navigation Arm
Number analyzed (Participants) | 26
participants
  Aspirating Needle: number analyzed (Participants) | 22
  Aspirating Needle | 15
  Biopsy Forcep: number analyzed (Participants) | 14
  Biopsy Forcep | 2
  Cytology Brush | 9
  superDimension Needle-Tipped Cytology Brush: number analyzed (Participants) | 2
  superDimension Needle-Tipped Cytology Brush | 2
  Gencut Core Biopsy Tool: number analyzed (Participants) | 5
  Gencut Core Biopsy Tool | 3
  superDimension Triple Needle Cytology Brush: number analyzed (Participants) | 1
  superDimension Triple Needle Cytology Brush | 1

15. Secondary Outcome: Diagnosis for Each Tool Based on Pathology of the ENB-aided Sample
Description: as for outcome 14
Time Frame: Based on final pathology results of the ENB-aided sample collected day of procedure
Population: Patients with overall malignant results by Pathology (30/49 cases). The number analyzed varies by tool based on the number of cases which used each tool. More than one tool could be used per case.
Measure: Number; unit: malignant results
Groups:
- Fluorscopic Navigation Arm: An Electromagnetic navigation bronchoscopy (ENB) system which provides enhanced three-dimensional fluoroscopy to improve lesion visibility and to compensate for CT-to-body divergence, with an integrated real-time local registration feature allowing the operator to update the catheter position relative to the target during the procedure.
Arm/Group | Fluorscopic Navigation Arm
Number analyzed (Participants) | 30
malignant results
  Aspirating Needle: number analyzed (Participants) | 25
  Aspirating Needle | 21
  Biopsy Forceps: number analyzed (Participants) | 16
  Biopsy Forceps | 12
  Cytology Brush | 20
  superDimension Needle-Tipped Cytology Brush: number analyzed (Participants) | 2
  superDimension Needle-Tipped Cytology Brush | 2
  Gencut Core Biopsy Tool: number analyzed (Participants) | 6
  Gencut Core Biopsy Tool | 5
  superDimension Triple Needle cytology Brush: number analyzed (Participants) | 1
  superDimension Triple Needle cytology Brush | 1
  Bronchoalveolar Lavage: number analyzed (Participants) | 16
  Bronchoalveolar Lavage | 10

16. Secondary Outcome: Percentage of Cases in Which the Intended Lesion is Correctly Identified
Description: In technically successful cases (local registration complete) the percentage of cases in which the intended lesion is correctly identified (as opposed to a non-target lesion or normal lung tissue) as indicated by the system software.
Time Frame: day of procedure
Population: 38 subjects had adequate video files to assess this endpoint
Measure: Count of Participants; unit: Participants
Arm/Group | Fluoroscopic Navigation Arm
Number analyzed (Participants) | 38
Participants
  correct identification of intended lesion | 38
  incorrect identification of intended lesion | 0

17. Secondary Outcome: Relational Accuracy in Cases in Which the Intended Lesion is Targeted
Description: In Technically successful cases (local registration complete) with evaluable videos the relational accuracy in cases in which the intended lesion is targeted was assessed. Relational accuracy is defined as the three-dimensional percentage overlap between the virtual target and the actual lesion in CBCT before (FNAV/CBCT 1) and after (FNAV/CBCT 2) correction of the catheter location.
Time Frame: day of procedure
Population: as for outcome 1
Measure: Median (Full Range); unit: 3D percent overlap
Arm/Group | Fluoroscopic Navigation Arm
Number analyzed (Participants) | 41
3D percent overlap
  Relational accuracy, Before location correction | 11.4 [0.0 to 97.0]
  Relational accuracy, after location correction | 32.8 [0.0 to 100.0]

ADVERSE EVENTS:
Time Frame: Adverse events will be collected after the ENB index procedure has been initiated (defined as introduction of the locatable guide or extended working channel into the subject). Adverse events will be collected immediately post procedure and at 7-day post procedure visit, with a window of 4-7 days post-procedure.
Description: An Adverse Event is any untoward medical occurrence, unintended disease or injury, or untoward clinical signs (including abnormal laboratory findings) in subjects, users or other persons, whether or not related to the investigational medical device.
  This definition includes events related to:
  1. the superDimension™ Navigation System v7.2 with Fluoroscopic Navigation Technology and all superDimension™ tools and accessories.
  2. the procedures involved, including bronchoscopy and sedation.
Arm/Group | Fluoroscopic Navigation Arm
All-Cause Mortality (participants affected / at risk) | 0/50
Serious Adverse Events (participants affected / at risk) | 1/50
Other Adverse Events (participants affected / at risk) | 7/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fluoroscopic Navigation Arm (N=50)
Infection (Infections and infestations) | 1 (1) — VIRAL ILLNESS
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fluoroscopic Navigation Arm (N=50)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 3 (3) — Coughing up blood
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Tiny left apical pneumothorax noted on post-bronchoscopic x-ray
Dizziness (Nervous system disorders) | 1 (1) — Patient feeling lightheaded, but it was relieved with rest.
Urinary Retention (Renal and urinary disorders) | 1 (1) — Difficulty urinating
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Chronic obstructive pulmonary disease (COPD) Exacerbation, shortness of breath

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institution/Investigator may publish the results of work performed under this Agreement, in accordance with the Publication Policy described in the Clinical Investigation Plan and publication guidelines from the Declaration of Helsinki. Institution and Investigator shall not publish the Study results until after Medtronic's Multi-site publication or until the elapse of twelve (12) months from the close of the Study at all Study sites, whichever occurs first.

DOCUMENTS (3):
  • Study Protocol: Clinical Investigation Plan (2018-04-09): https://cdn.clinicaltrials.gov/large-docs/59/NCT03585959/Prot_000.pdf
  • Statistical Analysis Plan (2019-05-21): https://cdn.clinicaltrials.gov/large-docs/59/NCT03585959/SAP_001.pdf
  • Study Protocol: Clinical Investigation Plan Note to File (2019-12-05): https://cdn.clinicaltrials.gov/large-docs/59/NCT03585959/Prot_002.pdf